CLINICAL TRIAL: NCT06692361
Title: Assessment of the Effectiveness and Safety of Fecal Microbiota Transplantation (FMT) in Patients With Major Depressive Disorder Who Do Not Show Early Improvement Following Antidepressant Treatment: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Assessment of the Efficacy and Safety of Fecal Microbiota Transplantation (FMT) in Patients With Major Depressive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gang Wang (Other)
Collaborators: Shandong Daizhuang Hospital (Unknown); Tianjin Anding Hospital (Other); The First Affiliated Hospital, Zhejiang University (Unknown); The First Hospital of Hebei Medical University (Other); West China Hospital (Other); Wuhu Fourth People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Gang Wang, Director of Beijing Anding Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No. 2024-58
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder (MDD); Depression - Major Depressive Disorder
Keywords: faecal microbiota transplantation; microbiome; major depressive disorder; RCT
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fecal Microbiota Transplantation; Microbiota; Escitalopram; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Escitalopram + FMT (Experimental): The experimental group will receive escitalopram + FMT capsules (using Oral capsules derived from healthy human fecal microbiota)
  Interventions: Biological: FMT capsule; Drug: Escitalopram (Lexapro)
- Escitalopram + placebo (Placebo Comparator): The control group will be treated with escitalopram + placebo (using capsules containing only corn starch)
  Interventions: Drug: Escitalopram (Lexapro); Biological: Corn Starch capsules

INTERVENTIONS:
Biological: FMT capsule — The experimental group will maintain escitalopram treatment and take 1.0 g of FMT capsules orally with breakfast every day for 4 weeks.
  Other Names: microbiota capsule; FMT
  Arms: Escitalopram + FMT
Drug: Escitalopram (Lexapro) — Both the experimental group and the placebo group were treated with the maximum tolerated dose of escitalopram.
  Other Names: Escitalopram
Biological: Corn Starch capsules — The placebo group will maintain escitalopram treatment and take corn starch capsules 1.0 g orally with breakfast every day for 4 weeks.
  Other Names: Corn starch
  Arms: Escitalopram + placebo

SUMMARY:
This study aimed to evaluate the efficacy and safety of fecal microbiota transplantation (FMT) in patients with major depressive disorder (MDD) who exhibit suboptimal early response to antidepressant treatment. Additionally, it sought to investigate the impact of FMT on biological indicators, including intestinal microbiota and metabolites, in individuals with MDD

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled study aims to compare the efficacy and safety of adjunctive FMT in patients with major depressive disorder (MDD) who show limited response to initial drug therapy.

A total of 600 patients experiencing depressive episodes will be screened, with all receiving escitalopram oxalate for an initial 2-week period. Of these, 214 participants who exhibit suboptimal therapeutic response to early antidepressant treatment will be enrolled and randomized in a 1:1 ratio to either the experimental group or control group.

During the intervention, participants will continue their existing antidepressant regimen and receive a 4-week treatment with either microbiota capsules or placebo. An additional 20-week follow-up assessment will then be conducted to evaluate outcomes.

ELIGIBILITY:
Inclusion Criteria (All 8 criterion are met):

* Outpatient or inpatient, aged 18 to 65 years (inclusive), regardless of gender;
* At the start of the screening phase, participants must meet the Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) diagnostic criteria for recurrent major depressive disorder (MDD) or single-episode MDD;
* At the start of the screening phase, participants' score on the 17-item Hamilton Depression Rating Scale (HAMD-17) must be ≥ 17;
* At the start of the screening phase, participants have not been treated with medication for their current depressive episode;
* At the start of the screening phase, participants are intended to be treated with a single antidepressant medication, Escitalopram;
* The HAMD-17 score after two weeks of treatment with the maximum tolerated dose of escitalopram was reduced by less than 20% compared with the HAMD-17 score at screening;
* Participants must have an education level above primary school and be able to understand the content of the scale;
* Participants sign the informed consent form.

Exclusion Criteria (Exclude if 1 criterion is met):

* According to DSM-5 criteria, currently or previously diagnosed as bipolar disorder, neurodevelopmental disorder, neurocognitive disorder, schizophrenia spectrum and other psychotic disorders, substance-related and addiction disorders;
* Accompanied by significant psychotic symptoms (delusions, hallucinations, etc.);
* The patient currently has severe or unstable central nervous system, cardiovascular, respiratory, liver, kidney, endocrine, blood system or other system diseases, and the researcher believes that the patient is not suitable for inclusion in this study;
* The patient currently has a serious suicide risk, and the HAMD-17 suicide risk item is ≥3 points;
* Suffering from inflammation-related diseases;
* Suffering from gastrointestinal infections, tumors and other structural abnormalities of the digestive system, including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease, etc.;
* Previous history of gastrointestinal surgery;
* Continuous use of antibiotics, probiotics, prebiotics or traditional Chinese medicine products for medical purposes for more than 2 weeks within 3 months before enrollment in the study;
* Those who are allergic to capsule ingredients and contents;
* Pregnant or lactating patients;
* Patients who are unable (such as difficulty swallowing) or unwilling to swallow capsules;
* Patients who received MECT treatment in the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The differences in efficacy(HAMD-17 score reduction rate ≥50%) between the two groups | Baseline, Week 4, Week 8
  The Hamilton Depression Rating Scale-17(HAMD-17) was used to assess the severity of depression in patients. If the HAMD-17 score reduction rate was ≥50%, the treatment was considered effective. 4 weeks after 4-week treatments, the differences in the effective rate of treatment between the two groups will be compared.

SECONDARY OUTCOMES:
The differences in complete remission rate(HAMD-17 ≤ 7 points) between the two groups | Baseline, Week 4, Week 8
  The Hamilton Depression Rating Scale-17 (HAMD-17) was used to assess the severity of depression in patients. 4 weeks after 4-week treatments, the differences in complete remission rate (HAMD-17 ≤ 7 points) between the two groups will be compared.
The differences in effective rate(HAMD-17 score reduction rate ≥50%) | Baseline and Week 4
  At the end of 4-week treatments, the differences in effective rate(HAMD-17 score reduction rate ≥ 50%) between the two groups will be compared.
The differences in complete remission rate(HAMD-17 ≤ 7 points) between the two groups | Baseline and Week 4
  At the end of 4-week treatments, the differences in complete remission rate(HAMD-17 ≤ 7 points) between the two groups will be compared.
Changes in total score of GAD-7 scale | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes in the total score of the Generalized Anxiety Disorder-7(GAD-7) scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes in total score of QIDS-SR scale | Baseline, Week 4, Week 8, Week 12, Week 24
  Quick Inventory of Depressive Symptoms-Self Rated(QIDS-SR) is mainly used to assess the severity of depressive symptoms. It includes 9 symptoms for depression diagnosis. QIDS-SR is very sensitive to changes in depressive symptoms. Changes in the total score of QIDS-SR scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
The differences in the reduction scores of the HAMD-17 scale in 4 symptom dimensions | Baseline, Week 4, Week 8, Week 12, Week 24
  The differences in the reduction scores of the HAMD-17 scale in 4 different symptom dimensions at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) was recorded: depression (1/2/3/7/8 items), anxiety (9/10/11/15/17 items), insomnia (4/5/6 items), and somatic (12/13/14/16 items).
Changes in total score of GSRS scale | Baseline, Week 4, Week 8, Week 12, Week 24
  The investigators will use the 7-level rating version of the Gastrointestinal Symptom Rating Scale(GSRS). Changes in the total score of the GSRS scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes in total score of SF-12 scale | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes in the total score of the Short Form 12 Health Survey(SF-12) scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes in total score of SDS scale | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes in the total score of the Sheehan Disability Scale(SDS) scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes in total score of PDQ-5D scale | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes in the total score of the Perceived Deficit Questionnaire for Depression 5-item(PDQ-5D) scale at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes of each subscale of CBCT | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes of each subscale of the Cognitive Behavioral Assessment Tool(CBCT) at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes of each subscale of CGI | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes of each subscale of the Clinical Global Impressions(CGI) at each follow-up time (0,4,8 and 20 weeks after 4-weeks treatments) will be compared with the total score at baseline.
Changes of each subscale of PSQI | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes of each subscale of the Pittsburgh sleep quality index(PSQI) at each follow-up time (0,4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Changes in brain imaging and EEG indicators | Baseline, Week 4, Week 8, Week 12, Week 24
  Changes in brain imaging and Electroencephalogram(EEG) indicators at each follow-up time (4,8 and 20 weeks after 4-week treatments) will be compared with the total score at baseline.
Evaluation of the safety of the treatments | Baseline, Week 4, Week 8, Week 12, Week 24
  The investigators will record any adverse events reported by participants, after treatments at each follow-up time (4,8 and 20 weeks after 4-week treatments).

OTHER OUTCOMES:
Explore changes in intestinal microbiota and metabolomics indicators related to FMT efficacy | Baseline, Week 4, Week 8, Week 12, Week 24
  Explore the changes in biological indicators at each follow-up time (0, 4, 8, and 20 weeks after 4-week treatments):
  1. Blood test: 1 procoagulant tube (5 ml), 1 PAXgene RNA collection tube (2.5 ml), 2 EDTA anticoagulant tubes (6 ml/tube);
  2. Urine test: 1 urine cup (40 ml);
  3. Feces test: 4 sets of feces samples and 2/3 of the 15 ml feces tube are used for microbiome, metabolome, proteome, transcriptome, epigenome and other omics detection and analysis.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Wuhu Fourth People's Hospital, Wuhu, Anhui
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Nangfang Hospital Affiliated of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Shandong Daizhuang Hospital, Jining, Shandong
  - West China Hospital Affiliated of Sichuan University, Chengdu, Sichuan
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali, Yunnan
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol